CLINICAL TRIAL: NCT02765100
Title: Depression, Obesity and Inflammatory Markers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Weill Cornell Medical College in Qatar (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1406015184
Record Dates: First submitted 2016-05-03; First posted 2016-05-06 (Estimated); Results first posted 2020-07-01 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Bipolar Disorder; Depression; Obesity
Keywords: Bipolar Disorder; Obesity; Depression
MeSH Terms: conditions — Bipolar Disorder; Depression; Obesity | interventions — Minocycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low CRP (Experimental): Subjects have CRP > 3
  Interventions: Drug: Minocycline
- High CRP (Experimental): Subjects have CRP =/> 3
  Interventions: Drug: Minocycline

INTERVENTIONS:
Drug: Minocycline — Minocycline 100 mg twice a day
  Other Names: Minocin

SUMMARY:
The purpose of this study is to better understand the relationship between bipolar disorder, body weight, and inflammation in the body (N=180). People with bipolar depression (N = 50)will be offered a place in a pilot study looking to see if the antibiotic minocycline added to current psychiatric medications has an effect on mood. A separate consent form will be provided for the pilot study. Numerous studies have documented the presence of altered immune function and elevation of inflammatory markers in patients with depression. Studies suggest that major depression is accompanied by immune dysregulation and activation of the inflammatory response system. While a small number of studies have found elevated inflammatory markers in bipolar mania, very little has been reported about inflammation in bipolar depression, and none of these studies have addressed the relationship of inflammatory markers with obesity in bipolar disorder.

DETAILED DESCRIPTION:
Aim 1 (N=180)will examine relationships between the levels of the inflammatory markers and current clinical state (depressed, manic or euthymic) with the hypothesis that Inflammatory markers will be higher in depression and mania relative to the euthymic state.

Aim 2 (N=180)will examine relationships between inflammatory markers and BMI in bipolar patients with the hypothesis that inflammatory markers will correlate positively with BMI.

Aim 3 (N=180)will examine the relationship between depression, obesity and inflammatory markers with the hypothesis that depressed (or manic) bipolar patients who are also obese will have higher inflammatory markers than either obese euthymic patients or non-obese depressed or manic patients.

Aim 4. (N=50) The pilot study will be to conduct a proof of concept add-on treatment study of the antibiotic minocycline for bipolar patients who are depressed, likely to be obese and likely to have elevated inflammatory markers and increased risk of heart disease. This is a proposal to conduct a 2-site trial of 50 subjects to examine the value of minocycline augmentation in bipolar depressed patients who are incompletely responsive to initial treatment with anti depressants and/or mood stabilizers. The investigators will compare two subgroups of depressed patients, those who have high (N=25) versus those who have low (N=25) levels of C-reactive protein (CRP).

ELIGIBILITY:
Inclusion Criteria:

* Patients with Bipolar Disorder and current depressive symptoms
* Hamilton Depression Scale score > 18
* Failed an adequate trial of at least one antidepressant or mood stabilizer of at least 4 weeks duration. Medication history will be recorded using the Antidepressant Treatment History Form
* 18 years or older
* Fluent in English or Arabic
* Have the capacity to understand the nature of the study and sign the written informed consent.

Exclusion Criteria:

* A current diagnosis of Schizophrenia or other psychotic disorder, or Dementia Alzheimer Type or related cognitive disorders.
* Principal diagnosis of Post-Traumatic Stress Disorder, Anorexia or Bulimia Nervosa, Obsessive-Compulsive Disorder. We define principal as the most pressing clinical problem.
* Pregnant or nursing
* Axis II diagnosis of antisocial, schizotypal or severe borderline personality disorder (defined as patients who are high risk for being unable to complete the study due to hospitalization, suicide attempts, significant self-mutilation, or other self-injurious or destructive behavior).
* Patients who currently meet criteria for Alcohol or other Substance-Related Dependence Disorder (with the exception of nicotine dependence) who require detoxification.
* Patients who are unable to read and write English or Arabic.
* Patients having serious, unstable or terminal medical or neurologic illness that would compromise study participation (i.e., metastatic or advanced malignancy, chronic renal failure requiring dialysis, recent myocardial infarction or unstable angina, or "end stage" chronic obstructive pulmonary disease). People with common conditions such as hypertension, insulin dependent diabetes mellitus, asthma, compensated congestive heart failure, a malignancy in remission, treated hypothyroidism, or epilepsy will not be excluded from participation.
* Autoimmune disease or chronic inflammatory diseases such as psoriasis or Crohn's disease
* Chronic infection such as hepatitis B or C or HIV
* Elevated antinuclear antibody or rheumatoid factor
* Oral glucocorticoids in the past 6 months
* Methotrexate or NSAID use in the past two weeks

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James H Kocsis, MD, Principal Investigator — Weill CMC
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared.

RESULTS

PARTICIPANT FLOW:
Groups:
- Low CRP: patients with a baseline C-ReactiveProtein value =/< 3 treated with minocycline 200 mg/d
- High CRP: patients with a baseline C-ReactiveProtein value >3 treated with minocycline 200 mg/d
Period: Overall Study
Arm/Group | Low CRP | High CRP
Started | 9 | 12
Completed | 8 | 10
Not Completed | 1 | 2
Not completed — subject found ineligible after baseline | 1 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Low CRP: CRP =/< 3
- High CRP: CRP > 3
- Total: Total of all reporting groups
Arm/Group | Low CRP | High CRP | Total
Number analyzed (Participants) | 9 | 12 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.3 (7.5) | 44.5 (14.0) | 48.3 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 9 | 11
  Male | 7 | 3 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 8 | 11 | 19
  Qatar | 1 | 1 | 2
Hamilton Depression Scale (HAMD) [Mean (Standard Deviation); unit: units on a scale] — Scores range from 0 (no depression) to 52 (most severe depression)
  units on a scale | 24.8 (6.5) | 23.0 (4.1) | 23.8 (5.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in Depression as Measured by the Hamilton Depression Scale Collected at Baseline and Week 8
Description: Scale ranges from 0-52. Greater change means greater improvement of depression from baseline to week 8.
Time Frame: Baseline; week 8
Population: Three participants not analyzed due to withdrawal from study
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Low CRP: patients with baseline CRP =/< 3
- High CRP: patients with baseline CRP > 3
Arm/Group | Low CRP | High CRP
Number analyzed (Participants) | 8 | 10
units on a scale | -12.2 (3.4) | -12.0 (3.1)
Statistical Analysis 1: Comparison: Low CRP vs High CRP; This is a pilot proof of concept study and does not require formal sample size calculations. High and low CRP groups will be compared on demographic, clinical and biological variables using two-sample t-tests or analysis of variance (ANOVA) tests for continuous variables (for nonparametric continuous variables, either Mann-Whitney tests or Kruskal-Wallis tests will be used) and chi-square tests or Fisher's exact tests for categorical variables; Test type: Equivalence — Unless specified otherwise, each of the statistical tests above will use a two-tailed alpha-level of 0.05; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = -0.2, Standard Deviation 3.4

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: Three participants not evaluated due to early withdrawal from the study
Arm/Group | Low CRP | High CRP
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/10
Other Adverse Events (participants affected / at risk) | 0/8 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-12): https://cdn.clinicaltrials.gov/large-docs/00/NCT02765100/Prot_SAP_000.pdf